CLINICAL TRIAL: NCT01403987
Title: Improving Performance of Paracentesis in Medical Residency Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Brian Jacobson, Associate Professor of Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: H-29983
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-09

CONDITIONS: Ascites; Cirrhosis
Keywords: Education; Ascites; Liver; Guidelines
MeSH Terms: conditions — Ascites; Fibrosis | interventions — Standard of Care; Audiovisual Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Arm (Active Comparator): Control group will receive standard teaching by the Residency Program regarding management of ascites and performance of paracentesis.
  Interventions: Behavioral: Residency Program Teaching
- Intermediate Education Arm (Experimental): In addition to the teaching provided by the residency program, the intermediate education group will receive a dedicated lecture by a gastroenterology fellow designed to teach consensus guidelines and their rationale in management of ascites. They will also receive a pocket card noting specific indications for paracentesis, and a brief summary of guidelines.
  Interventions: Behavioral: Residency Program Teaching; Behavioral: Lecture; Other: Pocket Card Reference
- Intensive Education Arm ("Pager" Arm) (Experimental): This group will receive the residency teaching, the specialist lecture, the pocket card, and have access to a pager carried by a gastroenterology fellow for personal assistance in performing paracentesis.
  Interventions: Behavioral: Residency Program Teaching; Behavioral: Lecture; Other: Pocket Card Reference; Behavioral: Pager

INTERVENTIONS:
Behavioral: Residency Program Teaching — The residency program provides education surrounding the management of ascites to all house-staff in the training program. This consists of lectures, case-based or bedside discussions, and board review. All arms will receive the standard teaching provided by the residency program.
  Other Names: Standard therapy
Behavioral: Lecture — During resident rotations on inpatient wards there are typically several dedicated, one-hour discussions facilitated by the team's supervising attending, addressing a variety of internal medicine topics. In place of or in addition to one of these discussions, a gastroenterology fellow will meet with the team for one hour to discuss a standardized case of a patient with ascites and the management issues. At this time they will review the consensus guidelines for management, and be provided with a pocket card with key points.
  Other Names: Didactic session
  Arms: Intensive Education Arm ("Pager" Arm); Intermediate Education Arm
Other: Pocket Card Reference — A 4x6 inch laminated card will be administered to both intervention arms at the beginning of the study. The card will contain a brief summary of AASLD guidelines, indications for and contraindications to paracentesis, and key studies to order for fluid analysis. The organization of residency rotations is such that members of one randomization group do not typically work with members of other groups, however in the event that there is crossover, they will be free to share information as they see fit in order to optimize patient care.
  Other Names: Visual aid
  Arms: Intensive Education Arm ("Pager" Arm); Intermediate Education Arm
Behavioral: Pager — The intensive education arm will be given a pager number at their initial meeting that they can use to call for personal assistance with performing paracentesis. Since a paracentesis is frequently referred to by housestaff as a "tap," the pager number will correlate with the letters, "TAPS," or #8277. The goal of the pager is to provide supervision and individual teaching so that the care provider can become proficient in the procedure.
  Other Names: One-on-one teaching
  Arms: Intensive Education Arm ("Pager" Arm)

SUMMARY:
The investigators hypothesize that there is significant variability in management of patients with ascites despite guidelines provided by the American Association for the Study of Liver Diseases, the professional organization most involved with management of liver patients. This variability may be attributable to knowledge deficits, skill limitations, or reflect systems-issues that limit the ability of a care provider to implement the clinical guidelines (time constraints, inadequate supervision, availability of appropriate equipment, and obtaining consent for non-emergent procedures). This variability does a disservice to the patients being treated, and results in trainee development of habits that are not evidence based. There are simple teaching tools available that may improve learning and retention of evidence based practice. Using these tools should result in more consistent appropriate patient care, improve patient outcomes, and provide better education to our trainees.

The purpose of this study is threefold: 1. To improve medical house-staff's technical performance of and comfort level with paracentesis; 2. To improve adherence to professional organization guidelines and to determine if this in fact improves clinical outcomes; 3. To evaluate efficacy of three teaching interventions in inpatient medicine trainee rotations.

DETAILED DESCRIPTION:
Since 2004 the American Association for the Study of Liver Disease (AASLD) has well-established guidelines for management of liver failure patients that is based on expert review of current literature. These guidelines address the initial evaluation of patients admitted to the hospital with complications of their liver disease, including patients with abdominal distention from fluid accumulation. In many cases, evaluation of this intraabdominal fluid, or ascites, performed using paracentesis, a procedure in which fluid is withdrawn from the abdomen and sent for laboratory analysis, is indicated, and the results of which will guide further treatment. Despite these guidelines, there remains significant variability in practice among inpatient providers.

The study will begin with a chart review to identify compliance with, and barriers to, evidence-based recommendations. A baseline survey of house-staff in the internal medicine department will be used to identify knowledge base and perceived barriers to implementation of best practices as defined by AASLD. The house-staff will subsequently be divided into three intervention groups for administration and evaluation of different teaching tools. A control group will have internet access to AASLD guidelines and undergo teaching that is already provided by the residency program. The second group will receive the baseline teaching, but also receive a pocket-card outlining recommendations and participate in a short, dedicated lecture to reinforce the guidelines. The third group will receive the pocket card, lecture, and a pager number to call for individual education at the time that cases arise. The groups will be followed for a period of six months, after which they will participate in an exit survey for reassessment of knowledge and perceived barriers, and a chart review will be conducted for comparison of data.

The primary outcome will be subjective improvement in practice based on survey results. Secondary outcomes will be measurement of actual and perceived benefit of pocket card, lecture, and individual education, determined by knowledge based questions on the survey, and improvement in patient clinical outcomes based on chart review noting particularly 30-day readmission rate and 90-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* All house-staff in the Internal Medicine Residency training program at Boston Medical Center; House-staff participating in Internal Medicine inpatient rotations as part of preliminary training for other specialties

Exclusion Criteria:

* House-staff participating in inpatient rotations not supervised by the Department of Internal Medicine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jacobson, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Runyon BA; AASLD Practice Guidelines Committee. Management of adult patients with ascites due to cirrhosis: an update. Hepatology. 2009 Jun;49(6):2087-107. doi: 10.1002/hep.22853. No abstract available. PMID 19475696
- [Background] Kashner TM, Henley SS, Golden RM, Byrne JM, Keitz SA, Cannon GW, Chang BK, Holland GJ, Aron DC, Muchmore EA, Wicker A, White H. Studying the effects of ACGME duty hours limits on resident satisfaction: results from VA learners' perceptions survey. Acad Med. 2010 Jul;85(7):1130-9. doi: 10.1097/ACM.0b013e3181e1d7e3. PMID 20592508
- [Background] Chahla M, Eberlein M, Wright S. The effect of providing a USB syllabus on resident reading of landmark articles. Med Educ Online. 2010 Jan 29;15. doi: 10.3402/meo.v15i0.4639. PMID 20165697
- [Background] Tomolo A, Caron A, Perz ML, Fultz T, Aron DC. The outcomes card. Development of a systems-based practice educational tool. J Gen Intern Med. 2005 Aug;20(8):769-71. doi: 10.1111/j.1525-1497.2005.0168.x. PMID 16050891
- [Background] Walton JM, Steinert Y. Patterns of interaction during rounds: implications for work-based learning. Med Educ. 2010 Jun;44(6):550-8. doi: 10.1111/j.1365-2923.2010.03626.x. PMID 20604851

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm | Intermediate Education Arm | Intensive Education Arm ("Pager" Arm)
Started | 34 | 34 | 68
Completed | 16 | 17 | 50
Not Completed | 18 | 17 | 18
Not completed — Residents forgot their secret PIN | 18 | 17 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Intermediate Education Arm | Intensive Education Arm ("Pager" Arm) | Total
Number analyzed (Participants) | 34 | 34 | 68 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 34 | 68 | 136
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: Number of participants] — Gender was not captured as a requirement of our IRB to limit ability to identify participants.
  Number of participants | NA — IRB would not allow capture of data | NA — IRB would not allow capture of data | NA — IRB would not allow capture of data | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68 | 136

OUTCOME MEASURES:

1. Primary Outcome: Score Out of Total Possible 25 on a Likert Scale.
Description: Primary outcome is quantified by summation of Likert scale responses to five questions assessing for comfort level in caring for and managing inpatients with ascites. The scale ranges from "strongly disagree," which is assigned a value of 1, to "strongly agree," assigned a value of 5. The summation scores will therefore range from 5 to 25 points out of a total of 25 possible points. The post-intervention scores will be compared between groups using a multiple regression model with terms for treatment, baseline summary scores, and other baseline demographic variables as needed.
Time Frame: 6 months
Population: Those who provided both baseline and follow up surveys
Measure: Mean (Standard Deviation); unit: units on a Likert scale (maximum is 25)
Arm/Group | Control Arm | Intermediate Education Arm | Intensive Education Arm ("Pager" Arm)
Number analyzed (Participants) | 16 | 17 | 50
units on a Likert scale (maximum is 25) | 21 (5) | 21 (5) | 20 (5)

2. Secondary Outcome: Improvement in Guideline Adherence
Description: Improvement in adherence to AASLD guidelines is summarized as yes or no improvement based on investigator chart review performed prior to and after the intervention. This is not a measure of resident reporting adherence but rather investigator interpretation of patient care and whether care was in line with published guidelines.
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Control Arm | Intermediate Education Arm | Intensive Education Arm ("Pager" Arm)
Number analyzed (Participants) | 16 | 17 | 50
percentage of participants | 44 | 53 | 80

3. Secondary Outcome: Readmission and Mortality Rates
Description: Percentage of patients in each arm that were either readmitted within 30 days or died within 90 days (ie a combined endpoint of either/or readmission or death)
Time Frame: 18 months
Measure: Number; unit: percentage of patients
Arm/Group | Control Arm | Intermediate Education Arm | Intensive Education Arm ("Pager" Arm)
Number analyzed (Participants) | 16 | 17 | 50
percentage of patients | 60 | 60 | 60

ADVERSE EVENTS:
Arm/Group | Control Arm | Intermediate Education Arm | Intensive Education Arm ("Pager" Arm)
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/68
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/68

LIMITATIONS AND CAVEATS:
Large number of participants lost to analysis because they forgot their secret personal ID number. The IRB had required we not have a way to link surveys to particular residents, and so lost power with loss of many residents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes